CLINICAL TRIAL: NCT00654771
Title: Prospective Comparison of Catheterized and Clean Catch Urine Specimens for Determination of Protein/Creatinine Ratio in Evaluation of Preeclampsia
Brief Title: Comparison of Catheterized and Clean Catch Urine Specimens for Protein/Creatinine Ratio in Preeclampsia Evaluation
Acronym: UPREE
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: Irene McLenahan Young Investigators Research Fund of the Magee-Womens Foundation (Unknown)
Responsible Party: Beatrice Chen
Other Study IDs: 0502110
Record Dates: First submitted 2008-04-03; First posted 2008-04-09 (Estimated); Last update posted 2012-08-16 (Estimated); Status verified 2012-08

CONDITIONS: Preeclampsia; Proteinuria; Hypertension; Pregnancy
Keywords: protein/creatinine ratio; clean catch urine; catheterized urine
MeSH Terms: conditions — Pre-Eclampsia; Proteinuria; Hypertension | interventions — Urine Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: women undergoing evaluation for pre-eclampsia
  Interventions: Other: urine collection

INTERVENTIONS:
Other: urine collection — clean catch urine collection and catheterized urine collection

SUMMARY:
The purpose of this prospective study was to examine whether protein/creatinine ratios in catheterized urine specimens correlate to clean catch specimens in pregnant patients being evaluated for preeclampsia.

DETAILED DESCRIPTION:
Preeclampsia is the new onset of hypertension and proteinuria after twenty weeks of gestation in pregnant women. The gold standard for evaluation of proteinuria in the diagnosis of preeclampsia is a twenty-four hour urine collection. However, single-specimen protein/creatinine ratios have been used to detect preeclampsia without the delay and inconvenience that a twenty-four hour urine collection would entail. At our institution, women are routinely catheterized for urine collection of protein/creatinine ratios because of concerns that vaginal contaminants would falsely elevate protein measurement in urine. However, no studies have specifically evaluated whether catheterized urine specimens correlate to clean catch urine specimens in protein estimation. Thus, the purpose of this prospective study was to examine whether protein/creatinine ratios in catheterized urine specimens correlate to clean catch specimens in pregnant patients being evaluated for preeclampsia.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant hypertensive patients between the ages of 14 - 50 of any gestational age greater than 20 weeks undergoing evaluation for preeclampsia

Exclusion Criteria:

* Ruptured membranes
* Any vaginal bleeding or spotting
* Pre-existing urinary tract infections or patients who are found to have a concurrent urinary tract infection upon culture of urine
* Patients who have previously been enrolled in the study

Ages: 14 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Any pregnant woman between the ages of 14 - 50 who is being evaluated for preeclampsia is eligible for this study.
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2005-07; Primary Completion 2006-05 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Correlation between protein/creatinine ratios for clean catch and catheterized urine specimens | time of enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Beatrice A Chen, MD, Principal Investigator — University of Pittsburgh Medical Center
Locations (1):
- Magee-Womens Hospital of UPMC, Pittsburgh, Pennsylvania, United States